CLINICAL TRIAL: NCT07118410
Title: Effect of Resistance Exercise With Blood Flow Restriction by Vascular Occlusion on Myocardial Function in Heart Failure With Reduced Ejection Fraction
Brief Title: Resistance Exercise With Blood Flow Restriction by Vascular Occlusion on Myocardial Function in Heart Failure With Reduced Ejection Fraction
Acronym: ERFOCARD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NIMAO/2024-2/CB-01
Record Dates: First submitted 2025-08-01; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Ventricular Function, Left
Keywords: Cardiac rehabilitation; Resistance training; Blood flow restriction; Cardiac function; Speckle tracking echography; Heart failure with reduced ejection fraction
MeSH Terms: conditions — Heart Failure | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups : blood flow restriction+resistance training group (BFR+RT) or the resistance training control group (RT). Patients will receive 4 weeks of cardiac rehabilitation with 6 sessions/week, 2 sessions of aerobic training on a cycloergometer and 4 sessions of RT with or without BFR depending on the group.
  Patients will be assessed at inclusion and at the end of the protocol by speckle tracking echocardiography, cardio-pulmonary test and muscular evaluation on isokinetic dynamometer.
Who Masked: Outcomes Assessor
Masking Description: The primary endpoint assessor is blinded to the group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT control group (No Intervention): Patients on resistance training only. Patients in this group will receive 4 weeks of cardiac rehabilitation with 6 sessions/week, 2 sessions of aerobic training on a cycloergometer and 4 sessions of resistance training
- RT+BFR group (Experimental): Patients on resistance training combined with blood flow restriction. Sessions will consist of 30 repetitions, followed by 3 sets of 15 repetitions at 40% 1-MR (maximal repetition), interspersed with 60 sec of recovery. An arterial occlusion pressure of 50% of systolic pressure will be maintained constant using a digital tourniquet. The cuff will be deflated during the recovery phases.
  Interventions: Device: Application of a vascular restriction device during resistance training

INTERVENTIONS:
Device: Application of a vascular restriction device during resistance training — In the BFR-RT group, sessions will consist of 30 repetitions, followed by 3 sets of 15 repetitions at 40% 1-MR (maximal repetition), interspersed with 60 sec of recovery. An arterial occlusion pressure of 50% of systolic pressure will be maintained constant using a digital tourniquet. The cuff will be deflated during the recovery phases.
  In the control group (RT group) it will be the same intervention with same intensities but without using BFR.
  Other Names: Resistance training
  Arms: RT+BFR group

SUMMARY:
Exercise is essential in cardiac rehabilitation for heart failure patients.Aerobic training and resistance training are both recommended. Resistance training improves muscle mass and strength and also improves the remodeling of cardiac function, thus reducing exercise intolerance in these patients. However, to obtain these adaptations, resistance training must be done at moderate to high intensities, which cannot always be sustained by the most fragile and deconditioned patients, such as those with reduced ejection fraction (Heart failure with reduced Ejection Fraction).

Blood flow restriction (BFR) by vascular occlusion training is an interesting alternative to conventional resistance training for these deconditioned patients. Preclinical and clinical studies have shown that, for low-intensity regimens, resistance training and blood flow restriction by vascular occlusion improves muscle strength and left ventricular function, unlike resistance training alone. Tissue hypoxemia, initiated by vascular occlusion and exacerbated by maintenance of exercise, is a key element in the peripheral adaptations documented in blood flow restriction, triggering a cascade of signaling pathways involving neurohumoral factors in particular, with effects both locally (i.e. striated skeletal muscle) and remotely, on the myocardium among others. The feasibility and safety of blood flow restriction in heart failure patients has been well demonstrated. Left ventricle ejection fraction remains a very global functional index, with poor reproducibility influenced by cardiac load conditions, making it impossible to draw any conclusions as to possible improvements in myocardial function, linked to changes in intrinsic tissue decontractility/relaxation properties. New cardiac imaging techniques like Speckle Tracking Echography have made it possible to assess the effects of blood flow resistance on myocardial function but so far no studies have used these tools to compare the effects of BFR+resistance training and resistance training alone on myocardial function in heart failure patients. It is suggested that resistance training combined with blood flow resistance could further improve cardiac and muscular function compared with resistance training alone, by activating neurohumoral mediators, like certain micro ribonucleic acids.

DETAILED DESCRIPTION:
Physical exercise is an essential part of cardiac rehabilitation for heart failure patients. In addition to aerobic training, resistance training is now recommended by scientific societies. Clinical studies report that resistance training contributes not only to peripheral reconditioning, with improved muscle mass and strength, but also to central reconditioning, with improved remodeling and cardiac function, thus reducing the exercise intolerance of heart failure patients. These favorable adaptations are achieved, however, on condition that RT is performed at moderate to high intensities (e.g. >75-80% of maximal repetition), intensities that cannot always be sustained by the most fragile and deconditioned patients, such as those with heart failure with reduced ejection fraction. The guidelines recommend intensities of 40% or less of repetition maximum.

Blood flow restriction (BFR) by vascular occlusion training is an interesting alternative to conventional resistance training, particularly for these most deconditioned patients. Preclinical and clinical studies have clearly established that for low-intensity regimens (around 40% of maximal repetition, an intensity well tolerated by the most fragile patients), resistance training+BFR improves muscle strength and left ventricular function, unlike resistance training alone. Tissue hypoxemia, initiated by vascular occlusion and exacerbated by maintenance of exercise, is a key element in the peripheral adaptations documented in BFR, triggering the activation of a cascade of signaling pathways involving neurohumoral factors in particular, with effects both locally (i.e. striated skeletal muscle) and remotely, on the myocardium among others. The feasibility and safety (i.e. no reported adverse events) of BFR in heart failure patients has been well demonstrated.

Left ventricular ejection fraction remains a very global functional index, with poor reproducibility and influenced by cardiac load conditions, making it impossible to draw any conclusions as to possible improvements in myocardial function, linked to changes in intrinsic tissue decontractility/relaxation properties. Innovative cardiac imaging techniques, such as Speckle Tracking Echography, now enable a detailed assessment of the effects of BFR on myocardial function. However, no study has yet used these tools to compare the effects of BFR+resistance training and resistance training alone on myocardial function in heart failure with reduced ejection patients. It is hypothetically suggested that resistance training combined with BFR could further improve cardiac and muscular function compared with resistance training alone, thanks to the activation of neurohumoral mediators, such as certain micro ribonucleic acids.

ELIGIBILITY:
Inclusion Criteria:

* LVEF ≤ 50%
* Patients with an indication for cardiovascular rehabilitation in the first stay or not (according to national recommendations, as soon as possible after an exacerbation or at any time in a patient with chronic heart failure) (Bigot et al., 2024)
* No medical contraindication to physical activity
* Patient has given free and informed consent and signed the consent form
* Patient affiliated with or benefiting from a health insurance scheme

Exclusion Criteria:

* Patient participating in another Category I interventional study, or having participated in another interventional study in the last month
* Patient in an exclusion period determined by a previous study
* Patient under court protection, guardianship or curatorship
* Unable to provide informed consent, or patient refuses to sign consent form
* Pregnant, parturient or breast-feeding patient
* Moderate to severe peripheral arterial disease. Arterial Doppler scan for arterial stenosis, with measurement of femoral and distal flows.
* Active or recent deep vein thrombosis. Check with venous Doppler ultrasound, looking for venous compressibility at the roots of the thighs, and 4-point venous ultrasound.
* Medication known to alter the effects of ischemic conditioning (cyclosporine, glibenclamide).
* Uncontrolled arterial hypertension
* Severe valvular disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
RT control group | Baseline
  Left ventricular global longitudinal strain (GLS), calculated from segmental longitudinal strains on apical 4-, 3-, and 2-chamber views using an 18-segment model (Voigt et al 2015).
BFR+RT group | Baseline
  Left ventricular global longitudinal strain (GLS), calculated from segmental longitudinal strains on apical 4-, 3-, and 2-chamber views using an 18-segment model (Voigt et al 2015).
RT control group | After 4 weeks of rehabilitation
  Left ventricular global longitudinal strain (GLS), calculated from segmental longitudinal strains on apical 4-, 3-, and 2-chamber views using an 18-segment model (Voigt et al 2015).
BFR+RT group | After 4 weeks of rehabilitation
  Left ventricular global longitudinal strain (GLS), calculated from segmental longitudinal strains on apical 4-, 3-, and 2-chamber views using an 18-segment model (Voigt et al 2015).

SECONDARY OUTCOMES:
(A) other parameters of left ventricular and atrial myocardial function in the control group: Myocardial work | Baseline
  The global index (constructive work, lost work, and efficiency) will be measured in mmHg%
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Myocardial work | Baseline
  The global index (constructive work, lost work, and efficiency) will be measured in mmHg%
(A) other parameters of left ventricular and atrial myocardial function in the control group: Myocardial work | After 4 weeks of rehabilitation
  The global index (constructive work, lost work, and efficiency) will be measured in mmHg%
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Myocardial work | After 4 weeks of rehabilitation
  The global index (constructive work, lost work, and efficiency) will be measured in mmHg%
(A) other parameters of left ventricular and atrial myocardial function in the control group: Left atrial deformities | Baseline
  Left atrial deformities will be measured in %
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Left atrial deformities | Baseline
  Left atrial deformities will be measured in %
(A) other parameters of left ventricular and atrial myocardial function in the control group: Left atrial deformities | After 4 weeks of rehabilitation
  Left atrial deformities will be measured in %
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Left atrial deformities | After 4 weeks of rehabilitation
  Left atrial deformities will be measured in %
(A) other parameters of left ventricular and atrial myocardial function in the control group: Mechanical dispersion | Baseline
  Post-systolic contractions will be measured in mmHg%
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Mechanical dispersion | Baseline
  Post-systolic contractions will be measured in mmHg%
(A) other parameters of left ventricular and atrial myocardial function in the control group: Mechanical dispersion | After 4 weeks of rehabilitation
  Post-systolic contractions will be measured in mmHg%
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Mechanical dispersion | After 4 weeks of rehabilitation
  Post-systolic contractions will be measured in mmHg%
(A) other parameters of left ventricular and atrial myocardial function in the control group: Left ventricle ejection fraction | Baseline
  Left ventricle ejection fraction will be measured in %
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Left ventricle ejection fraction | Baseline
  Left ventricle ejection fraction will be measured in %
(A) other parameters of left ventricular and atrial myocardial function in the control group: Left ventricle ejection fraction | After 4 weeks of rehabilitation
  Left ventricle ejection fraction will be measured in %
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Left ventricle ejection fraction | After 4 weeks of rehabilitation
  Left ventricle ejection fraction will be measured in %
(A) other parameters of left ventricular and atrial myocardial function in the control group: E/E' and E/A ratio | Baseline
  E/E' and E/A ratio will be measured
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: E/E' and E/A ratio | Baseline
  E/E' and E/A ratio will be measured
(A) other parameters of left ventricular and atrial myocardial function in the control group: E/E' and E/A ratio | After 4 weeks of rehabilitation
  E/E' and E/A ratio will be measured
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RTgroup: E/E' and E/A ratio | After 4 weeks of rehabilitation
  E/E' and E/A ratio will be measured
(A) other parameters of left ventricular and atrial myocardial function in the control group: Cardiac index | Baseline
  Cardiac index will be measured in L/min/m2
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Cardiac index | Baseline
  Cardiac index will be measured in L/min/m2
(A) other parameters of left ventricular and atrial myocardial function in the control group: Cardiac index | After 4 weeks of rehabilitation
  Cardiac index will be measured in L/min/m2
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Cardiac index | After 4 weeks of rehabilitation
  Cardiac index will be measured in L/min/m2
(A) other parameters of left ventricular and atrial myocardial function in the control group: Tricuspid regurgitation flow | Baseline
  Tricuspid regurgitation flow will be measured in m/sec
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Tricuspid regurgitation flow | Baseline
  Tricuspid regurgitation flow will be measured in m/sec
(A) other parameters of left ventricular and atrial myocardial function in the control group: Tricuspid regurgitation flow | After 4 weeks of rehabilitation
  Tricuspid regurgitation flow will be measured in m/sec
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Tricuspid regurgitation flow | After 4 weeks of rehabilitation
  Tricuspid regurgitation flow will be measured in m/sec
(A) other parameters of left ventricular and atrial myocardial function in the control group: systolic pulmonary arterial pressure | Baseline
  Systolic pulmonary arterial pressure will be measured in mmHg
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: systolic pulmonary arterial pressure | Baseline
  Systolic pulmonary arterial pressure will be measured in mmHg
(A) other parameters of left ventricular and atrial myocardial function in the control group: systolic pulmonary arterial pressure (mmHg) | After 4 weeks of rehabilitation
  Systolic pulmonary arterial pressure will be measured in mmHg
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: systolic pulmonary arterial pressure (mmHg) | After 4 weeks of rehabilitation
  Systolic pulmonary arterial pressure will be measured in mmHg
(A) other parameters of left ventricular and atrial myocardial function in the control group: Vmax IT | Baseline
  Vmax IT will be measured in m/sec
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Vmax IT | Baseline
  Vmax IT will be measured in m/sec
(A) other parameters of left ventricular and atrial myocardial function in the control group: Vmax IT | After 4 weeks of rehabilitation
  Vmax IT will be measured in m/sec
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Vmax IT | After 4 weeks of rehabilitation
  Vmax IT will be measured in m/sec
(A) other parameters of left ventricular and atrial myocardial function in the control group: Left ventricular volume | Baseline
  Left ventricular telesystolic and telediastolic volumes will be measured
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Left ventricular volume | Baseline
  Left ventricular telesystolic and telediastolic volumes will be measured
(A) other parameters of left ventricular and atrial myocardial function in the control group: Left ventricular volume | After 4 weeks of rehabilitation
  Left ventricular telesystolic and telediastolic volumes will be measured
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Left ventricular volume | After 4 weeks of rehabilitation
  Left ventricular telesystolic and telediastolic volumes will be measured
(A) other parameters of left ventricular and atrial myocardial function in the control group: Atrial volume | Baseline
  Atrial telesystolic and telediastolic volumes will be measured
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Atrial volume | Baseline
  Atrial telesystolic and telediastolic volumes will be measured
(A) other parameters of left ventricular and atrial myocardial function in the control group: Atrial volume | After 4 weeks of rehabilitation
  Atrial telesystolic and telediastolic volumes will be measured
(A) other parameters of left ventricular and atrial myocardial function in the BFR+RT group: Atrial volume | After 4 weeks of rehabilitation
  Atrial telesystolic and telediastolic volumes will be measured
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Myocardial work | Baseline
  The global index (constructive work, lost work, and efficiency) will be measured in mmHg%
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Myocardial work | Baseline
  The global index (constructive work, lost work, and efficiency) will be measured in mmHg%
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Myocardial work | After 4 weeks of rehabilitation
  The global index (constructive work, lost work, and efficiency) will be measured in mmHg%
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Myocardial work | After 4 weeks of rehabilitation
  The global index (constructive work, lost work, and efficiency) will be measured in mmHg%
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Left atrial deformities | Baseline
  Left atrial deformities will be measured in %
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Left atrial deformities | Baseline
  Left atrial deformities will be measured in %
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Left atrial deformities | After 4 weeks of rehabilitation
  Left atrial deformities will be measured in %
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Left atrial deformities | After 4 weeks of rehabilitation
  Left atrial deformities will be measured in %
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Mechanical dispersion | Baseline
  Post-systolic contractions will be measured in mmHg%
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Mechanical dispersion | Baseline
  Post-systolic contractions will be measured in mmHg%
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Mechanical dispersion | After 4 weeks of rehabilitation
  Post-systolic contractions will be measured in mmHg%
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Mechanical dispersion | After 4 weeks of rehabilitation
  Post-systolic contractions will be measured in mmHg%
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Left ventricle ejection fraction | Baseline
  The left ventricle ejection fraction will be measured as a percentage
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Left ventricle ejection fraction | Baseline
  The left ventricle ejection fraction will be measured as a percentage
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Left ventricle ejection fraction | After 4 weeks of rehabilitation
  The left ventricle ejection fraction will be measured as a percentage
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Left ventricle ejection fraction | After 4 weeks of rehabilitation
  The left ventricle ejection fraction will be measured as a percentage
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: E/E' and E/A ratio | Baseline
  The E/E' and E/A ratio will be measured
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: E/E' and E/A ratio | Baseline
  The E/E' and E/A ratio will be measured
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: E/E' and E/A ratio | After 4 weeks of rehabilitation
  The E/E' and E/A ratio will be measured
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: E/E' and E/A ratio | After 4 weeks of rehabilitation
  The E/E' and E/A ratio will be measured
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: cardiac index | Baseline
  Cardiac index will be measured in L/min/m2
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: cardiac index | Baseline
  Cardiac index will be measured in L/min/m2
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: cardiac index | After 4 weeks of rehabilitation
  Cardiac index will be measured in L/min/m2
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: cardiac index | After 4 weeks of rehabilitation
  Cardiac index will be measured in L/min/m2
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Tricuspid regurgitation flow | Baseline
  Tricuspid regurgitation flow will be measured in m/sec
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Tricuspid regurgitation flow | Baseline
  Tricuspid regurgitation flow will be measured in m/sec
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Tricuspid regurgitation flow | After 4 weeks of rehabilitation
  Tricuspid regurgitation flow will be measured in m/sec
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Tricuspid regurgitation flow | After 4 weeks of rehabilitation
  Tricuspid regurgitation flow will be measured in m/sec
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: systolic pulmonary arterial pressure | Baseline
  Systolic pulmonary arterial pressure will be measured in mmHg
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: systolic pulmonary arterial pressure | Baseline
  Systolic pulmonary arterial pressure will be measured in mmHg
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: systolic pulmonary arterial pressure | After 4 weeks of rehabilitation
  Systolic pulmonary arterial pressure will be measured in mmHg
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: systolic pulmonary arterial pressure | After 4 weeks of rehabilitation
  Systolic pulmonary arterial pressure will be measured in mmHg
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Vmax IT | Baseline
  Vmax IT will be measured in m/sec
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Vmax IT | Baseline
  Vmax IT will be measured in m/sec
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Vmax IT | After 4 weeks of rehabilitation
  Vmax IT will be measured in m/sec
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Vmax IT | After 4 weeks of rehabilitation
  Vmax IT will be measured in m/sec
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Atrial volume | Baseline
  Atrial telesystolic and telediastolic volumes will be measured
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Atrial volume | Baseline
  Atrial telesystolic and telediastolic volumes will be measured
(B) Left cardiac remodeling (left ventricle and atrium) in the control group: Atrial volume | After 4 weeks of rehabilitation
  Atrial telesystolic and telediastolic volumes will be measured
(B) Left cardiac remodeling (left ventricle and atrium) in the BFR+RT group: Atrial volume | After 4 weeks of rehabilitation
  Atrial telesystolic and telediastolic volumes will be measured
(C) Stress test measurement in controls : peak oxygen consumption | Baseline
  Peak oxygen consumption (VO2pic) will be measured in mL/min/kg
(C) Stress test measurement in the BFR+RT group : peak oxygen consumption | Baseline
  Peak oxygen consumption (VO2pic) will be measured in mL/min/kg
(C) Stress test measurement in controls : peak oxygen consumption | After 4 weeks of rehabilitation
  Peak oxygen consumption (VO2pic) will be measured in mL/min/kg
(C) Stress test measurement in the BFR+RT group: peak oxygen consumption | After 4 weeks of rehabilitation
  Peak oxygen consumption (VO2pic) will be measured in mL/min/kg
(C) Stress test measurement in controls : Maximum aerobic power | Baseline
  Maximum aerobic power will be measured in Watts
  * First ventilatory threshold (SV1) mL/min/kg
(C) Stress test measurement in the BFR+RT group : Maximum aerobic power | Baseline
  Maximum aerobic power will be measured in Watts
  * First ventilatory threshold (SV1) mL/min/kg
(C) Stress test measurement in controls : Maximum aerobic power | After 4 weeks of rehabilitation
  Maximum aerobic power will be measured in Watts
  * First ventilatory threshold (SV1) mL/min/kg
(C) Stress test measurement in the BFR+RT group : Maximum aerobic power | After 4 weeks of rehabilitation
  Maximum aerobic power will be measured in Watts
  * First ventilatory threshold (SV1) mL/min/kg
(C) Stress test measurement in controls : First ventilatory threshold | Baseline
  First ventilatory threshold will be measured in mL/min/kg
(C) Stress test measurement in the BFR+RT group : First ventilatory threshold | Baseline
  First ventilatory threshold will be measured in mL/min/kg
(C) Stress test measurement in controls : First ventilatory threshold | After 4 weeks of rehabilitation
  First ventilatory threshold will be measured in mL/min/kg
(C) Stress test measurement in the BFR+RT group : First ventilatory threshold | After 4 weeks of rehabilitation
  First ventilatory threshold will be measured in mL/min/kg
(C) Muscular evaluation in controls: Peak torque | Baseline
  Peak torque will be measured in Nm
(C) Muscular evaluation in the BFR+RT group: Peak torque | Baseline
  Peak torque will be measured in Nm
(C) Muscular evaluation in controls: Peak torque | After 4 weeks of rehabilitation
  Peak torque will be measured in Nm
(C) Muscular evaluation in the BFR+RT group: Peak torque | After 4 weeks of rehabilitation
  Peak torque will be measured in Nm
(C) Muscular evaluation in controls: Maximum repetition | Baseline
  Maximum repetition will be measured in kilograms
(C) Muscular evaluation in the BFR+RT group: Maximum repetition | Baseline
  Maximum repetition will be measured in kilograms
(C) Muscular evaluation in controls: Maximum repetition | After 4 weeks of rehabilitation
  Maximum repetition will be measured in kilograms
(C) Muscular evaluation in the BFR+RT group: Maximum repetition | After 4 weeks of rehabilitation
  Maximum repetition will be measured in kilograms
(D) Clinical and biological measurement in controls: Body mass index | Baseline
  Body mass index will be measured in Kg/m2
(D) Clinical and biological measurement in the BFR+RT group: Body mass index | Baseline
  Body mass index will be measured in Kg/m2
(D) Clinical and biological measurement in controls: Body mass index | After 4 weeks of rehabilitation
  Body mass index will be measured in Kg/m2
(D) Clinical and biological measurement in the BFR+RT group: Body mass index | After 4 weeks of rehabilitation
  Body mass index will be measured in Kg/m2
(D) Clinical and biological measurement in controls: Waist circumference | Baseline
  Waist circumference will be measured in cm
(D) Clinical and biological measurement in the BFR+RT group: Waist circumference | Baseline
  Waist circumference will be measured in cm
(D) Clinical and biological measurement in controls: Waist circumference | After 4 weeks of rehabilitation
  Waist circumference will be measured in cm
(D) Clinical and biological measurement in the BFR+RT group: Waist circumference | After 4 weeks of rehabilitation
  Waist circumference will be measured in cm
(D) Clinical and biological measurement in controls: Lipid profile | Baseline
  Lipids will be measured in mmol/L
(D) Clinical and biological measurement in the BFR+RT group: Lipid profile | Baseline
  Lipids will be measured in mmol/L
(D) Clinical and biological measurement in controls: Lipid profile | After 4 weeks of rehabilitation
  Lipids will be measured in mmol/L
(D) Clinical and biological measurement in the BFR+RT group: Lipid profile | After 4 weeks of rehabilitation
  Lipids will be measured in mmol/L
(D) Clinical and biological measurement in controls: Glycated hemoglobin | Baseline
  Glycated hemoglobin will be measured as a %
(D) Clinical and biological measurement in the BFR+RT group: Glycated hemoglobin | Baseline
  Glycated hemoglobin will be measured as a %
(D) Clinical and biological measurement in controls: Glycated hemoglobin | After 4 weeks of rehabilitation
  Glycated hemoglobin will be measured as a %
(D) Clinical and biological measurement in the BFR+RT group: Glycated hemoglobin | After 4 weeks of rehabilitation
  Glycated hemoglobin will be measured as a %
(D) Clinical and biological measurement in controls: Fasting blood glucose | Baseline
  Fasting blood glucose will be measured in g/L
(D) Clinical and biological measurement in the BFR+RT group: Fasting blood glucose | Baseline
  Fasting blood glucose will be measured in g/L
(D) Clinical and biological measurement in controls: Fasting blood glucose | After 4 weeks of rehabilitation
  Fasting blood glucose will be measured in g/L
(D) Clinical and biological measurement in the BFR+RT group: Fasting blood glucose | After 4 weeks of rehabilitation
  Fasting blood glucose will be measured in g/L
(D) Clinical and biological measurement in controls: Pro-Brain Natriuretic Peptide | Baseline
  Pro-Brain Natriuretic Peptide will be measured in ng/L
(D) Clinical and biological measurement in the BFR+RT group: Pro-Brain Natriuretic Peptide | Baseline
  Pro-Brain Natriuretic Peptide will be measured in ng/L
(D) Clinical and biological measurement in controls: Pro-Brain Natriuretic Peptide | After 4 weeks of rehabilitation
  Pro-Brain Natriuretic Peptide will be measured in ng/L
(D) Clinical and biological measurement in the BFR+RT group: Pro-Brain Natriuretic Peptide | After 4 weeks of rehabilitation
  Pro-Brain Natriuretic Peptide will be measured in ng/L
(D) Clinical and biological measurement in controls: C-reactive protein | Baseline
  C-reactive protein will be measured in mg/L
(D) Clinical and biological measurement in the BFR+RT group: C-reactive protein | Baseline
  C-reactive protein will be measured in mg/L
(D) Clinical and biological measurement in controls: C-reactive protein | After 4 weeks of rehabilitation
  C-reactive protein will be measured in mg/L
(D) Clinical and biological measurement in the BFR+RT group: C-reactive protein | After 4 weeks of rehabilitation
  C-reactive protein will be measured in mg/L
(D) Clinical and biological measurement in controls: Micro ribonucleic acids | Baseline
  Micro ribonucleic acids will be measured in ng/µl
(D) Clinical and biological measurement in the BFR+RT group: Micro ribonucleic acids | Baseline
  Micro ribonucleic acids will be measured in ng/µl
(D) Clinical and biological measurement in controls: Micro ribonucleic acid | After 4 weeks of rehabilitation
  Micro ribonucleic acids will be measured in ng/µl
(D) Clinical and biological measurement in the BFR+RT group: Micro ribonucleic acid | After 4 weeks of rehabilitation
  Micro ribonucleic acids will be measured in ng/µl
(E) MacNew Heart Disease Quality of Life score in controls | Baseline
  The MacNew is a self-administered heart disease-specific health-related quality of life [HRQL] questionnaire which addresses 3 major HRQL domains: Emotional, Physical, and Social. Each domain contains 9 questions to be rated as 1 [not very important] to 5 [very important]. These domains can be combined to give a Global HRQL score
(E) MacNew Heart Disease Quality of Life score in the BFR+RT group | Baseline
  The MacNew is a self-administered heart disease-specific health-related quality of life [HRQL] questionnaire which addresses 3 major HRQL domains: Emotional, Physical, and Social. Each domain contains 9 questions to be rated as 1 [not very important] to 5 [very important]. These domains can be combined to give a Global HRQL score
(E) MacNew Heart Disease Quality of Life score in controls | After 4 weeks of rehabilitation
  The MacNew is a self-administered heart disease-specific health-related quality of life [HRQL] questionnaire which addresses 3 major HRQL domains: Emotional, Physical, and Social. Each domain contains 9 questions to be rated as 1 [not very important] to 5 [very important]. These domains can be combined to give a Global HRQL score
(E) MacNew Heart Disease Quality of Life score in the BFR+RT group | After 4 weeks of rehabilitation
  The MacNew is a self-administered heart disease-specific health-related quality of life [HRQL] questionnaire which addresses 3 major HRQL domains: Emotional, Physical, and Social. Each domain contains 9 questions to be rated as 1 [not very important] to 5 [very important]. These domains can be combined to give a Global HRQL score
(F) International Physical Activity Questionnaire in controls | Baseline
  The International Physical Activity Questionnaire is intended for people aged 15 and over. The questionnaire assesses overall physical activity and sedentary time over the last seven days. The questionnaire looks at vigorous and moderate activity, walking, and time spent sitting (sedentary lifestyle), whether during leisure activities, at work, in daily life or during transport. There are several versions of the questionnaire, including a short one (7 questions) and a long one (27 questions), which people can self-administer or answer by telephone, for example. The questionnaire classifies the subject according to 3 levels of activity: inactive, moderate, high.
(F) International Physical Activity Questionnaire in the BFR+RT group | Baseline
  The International Physical Activity Questionnaire is intended for people aged 15 and over. The questionnaire assesses overall physical activity and sedentary time over the last seven days. The questionnaire looks at vigorous and moderate activity, walking, and time spent sitting (sedentary lifestyle), whether during leisure activities, at work, in daily life or during transport. There are several versions of the questionnaire, including a short one (7 questions) and a long one (27 questions), which people can self-administer or answer by telephone, for example. The questionnaire classifies the subject according to 3 levels of activity: inactive, moderate, high.
(F) International Physical Activity Questionnaire in controls | After 4 weeks of rehabilitation
  The International Physical Activity Questionnaire is intended for people aged 15 and over. The questionnaire assesses overall physical activity and sedentary time over the last seven days. The questionnaire looks at vigorous and moderate activity, walking, and time spent sitting (sedentary lifestyle), whether during leisure activities, at work, in daily life or during transport. There are several versions of the questionnaire, including a short one (7 questions) and a long one (27 questions), which people can self-administer or answer by telephone, for example. The questionnaire classifies the subject according to 3 levels of activity: inactive, moderate, high.
(F) International Physical Activity Questionnaire in the BFR+RT group | After 4 weeks of rehabilitation
  The International Physical Activity Questionnaire is intended for people aged 15 and over. The questionnaire assesses overall physical activity and sedentary time over the last seven days. The questionnaire looks at vigorous and moderate activity, walking, and time spent sitting (sedentary lifestyle), whether during leisure activities, at work, in daily life or during transport. There are several versions of the questionnaire, including a short one (7 questions) and a long one (27 questions), which people can self-administer or answer by telephone, for example. The questionnaire classifies the subject according to 3 levels of activity: inactive, moderate, high.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle ROBERT, Dr., Study Director — Nîmes University Hospital; Alice GAUTHIER, Dr., Principal Investigator — Nîmes University Hospital; Clara GROMOFF, Dr., Principal Investigator — Nîmes University Hospital; Bertrand LEDERMANN, Dr., Principal Investigator — Nîmes University Hospital; Philippe OBERT, Dr., Principal Investigator — UFR Sciences Technologies Centre INRAE, Avignon
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France

REFERENCES:
- [Background] Ambrosetti M, Abreu A, Corra U, Davos CH, Hansen D, Frederix I, Iliou MC, Pedretti RFE, Schmid JP, Vigorito C, Voller H, Wilhelm M, Piepoli MF, Bjarnason-Wehrens B, Berger T, Cohen-Solal A, Cornelissen V, Dendale P, Doehner W, Gaita D, Gevaert AB, Kemps H, Kraenkel N, Laukkanen J, Mendes M, Niebauer J, Simonenko M, Zwisler AO. Secondary prevention through comprehensive cardiovascular rehabilitation: From knowledge to implementation. 2020 update. A position paper from the Secondary Prevention and Rehabilitation Section of the European Association of Preventive Cardiology. Eur J Prev Cardiol. 2021 May 14;28(5):460-495. doi: 10.1177/2047487320913379. PMID 33611446
- [Background] Badano LP, Kolias TJ, Muraru D, Abraham TP, Aurigemma G, Edvardsen T, D'Hooge J, Donal E, Fraser AG, Marwick T, Mertens L, Popescu BA, Sengupta PP, Lancellotti P, Thomas JD, Voigt JU; Industry representatives; Reviewers: This document was reviewed by members of the 2016-2018 EACVI Scientific Documents Committee. Standardization of left atrial, right ventricular, and right atrial deformation imaging using two-dimensional speckle tracking echocardiography: a consensus document of the EACVI/ASE/Industry Task Force to standardize deformation imaging. Eur Heart J Cardiovasc Imaging. 2018 Jun 1;19(6):591-600. doi: 10.1093/ehjci/jey042. PMID 29596561
- [Background] Beckers PJ, Denollet J, Possemiers NM, Wuyts FL, Vrints CJ, Conraads VM. Combined endurance-resistance training vs. endurance training in patients with chronic heart failure: a prospective randomized study. Eur Heart J. 2008 Aug;29(15):1858-66. doi: 10.1093/eurheartj/ehn222. Epub 2008 May 30. PMID 18515805
- [Background] Bigot M, Guy JM, Monpere C, Cohen-Solal A, Pavy B, Iliou MC, Bosser G, Corone S, Douard H, Farrokhi T, Guerder A, Guillo P, Houppe JP, Pezel T, Pierre B, Roueff S, Thomas D, Verges B, Blanchard JC, Ghannem M, Marcadet D. Cardiac rehabilitation recommendations of the Group Exercise Rehabilitation Sports - Prevention (GERS-P) of the French Society of Cardiology: 2023 update. Arch Cardiovasc Dis. 2024 Aug-Sep;117(8-9):521-541. doi: 10.1016/j.acvd.2024.05.119. Epub 2024 Jul 4. No abstract available. PMID 39174436
- [Background] Billah M, Ridiandries A, Allahwala U, Mudaliar H, Dona A, Hunyor S, Khachigian LM, Bhindi R. Circulating mediators of remote ischemic preconditioning: search for the missing link between non-lethal ischemia and cardioprotection. Oncotarget. 2019 Jan 4;10(2):216-244. doi: 10.18632/oncotarget.26537. eCollection 2019 Jan 4. PMID 30719216
- [Background] Birnbaum Y, Hale SL, Kloner RA. Ischemic preconditioning at a distance: reduction of myocardial infarct size by partial reduction of blood supply combined with rapid stimulation of the gastrocnemius muscle in the rabbit. Circulation. 1997 Sep 2;96(5):1641-6. doi: 10.1161/01.cir.96.5.1641. PMID 9315559
- [Background] Botker HE, Lassen TR, Jespersen NR. Clinical translation of myocardial conditioning. Am J Physiol Heart Circ Physiol. 2018 Jun 1;314(6):H1225-H1252. doi: 10.1152/ajpheart.00027.2018. Epub 2018 Mar 2. PMID 29498531
- [Background] Cahalin LP, Formiga MF, Owens J, Anderson B, Hughes L. Beneficial Role of Blood Flow Restriction Exercise in Heart Disease and Heart Failure Using the Muscle Hypothesis of Chronic Heart Failure and a Growing Literature. Front Physiol. 2022 Jul 6;13:924557. doi: 10.3389/fphys.2022.924557. eCollection 2022. PMID 35874535
- [Background] Caminiti G, Volterrani M, Iellamo F, Marazzi G, Silvestrini M, Giamundo DM, Morsella V, Di Biasio D, Franchini A, Perrone MA. Exercise training for patients with heart failure and preserved ejection fraction. A narrative review. Monaldi Arch Chest Dis. 2025 Oct 14;95(3). doi: 10.4081/monaldi.2024.3030. Epub 2024 Jul 23. PMID 39058025
- [Background] Chen YC, Chen WC, Liu CW, Huang WY, Lu I, Lin CW, Huang RY, Chen JS, Huang CH. Is moderate resistance training adequate for older adults with sarcopenia? A systematic review and network meta-analysis of RCTs. Eur Rev Aging Phys Act. 2023 Nov 29;20(1):22. doi: 10.1186/s11556-023-00333-4. PMID 38030985
- [Background] Danduboyina A, Panjiyar BK, Borra SR, Panicker SS. Cardiovascular Benefits of Resistance Training in Patients With Heart Failure With Reduced Ejection Fraction: A Systematic Review. Cureus. 2023 Oct 27;15(10):e47813. doi: 10.7759/cureus.47813. eCollection 2023 Oct. PMID 38021681
- [Background] Eser P, Trachsel LD, Marcin T, Herzig D, Freiburghaus I, De Marchi S, Zimmermann AJ, Schmid JP, Wilhelm M. Short- and Long-Term Effects of High-Intensity Interval Training vs. Moderate-Intensity Continuous Training on Left Ventricular Remodeling in Patients Early After ST-Segment Elevation Myocardial Infarction-The HIIT-EARLY Randomized Controlled Trial. Front Cardiovasc Med. 2022 Jun 17;9:869501. doi: 10.3389/fcvm.2022.869501. eCollection 2022. PMID 35783836
- [Background] Fayol A, Wack M, Livrozet M, Carves JB, Domenge O, Vermersch E, Mirabel M, Karras A, Le Guen J, Blanchard A, Azizi M, Amar L, Bories MC, Mousseaux E, Carette C, Puymirat E, Hagege A, Jannot AS, Hulot JS. Aetiological classification and prognosis in patients with heart failure with preserved ejection fraction. ESC Heart Fail. 2022 Feb;9(1):519-530. doi: 10.1002/ehf2.13717. Epub 2021 Nov 29. PMID 34841727
- [Background] Ferraz RB, Gualano B, Rodrigues R, Kurimori CO, Fuller R, Lima FR, DE Sa-Pinto AL, Roschel H. Benefits of Resistance Training with Blood Flow Restriction in Knee Osteoarthritis. Med Sci Sports Exerc. 2018 May;50(5):897-905. doi: 10.1249/MSS.0000000000001530. PMID 29266093
- [Background] Junior AF, Schamne JC, Perandini LAB, Chimin P, Okuno NM. Effects of Walking Training with Restricted Blood Flow on HR and HRV Kinetics and HRV Recovery. Int J Sports Med. 2019 Sep;40(9):585-591. doi: 10.1055/a-0942-7479. Epub 2019 Jul 4. PMID 31272111
- [Background] Kambic T, Jug B, Piepoli MF, Lainscak M. Is blood flow restriction resistance training the missing piece in cardiac rehabilitation of frail patients? Eur J Prev Cardiol. 2023 Jan 24;30(2):117-122. doi: 10.1093/eurjpc/zwac048. No abstract available. PMID 35253869
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077
- [Background] Long L, Mordi IR, Bridges C, Sagar VA, Davies EJ, Coats AJ, Dalal H, Rees K, Singh SJ, Taylor RS. Exercise-based cardiac rehabilitation for adults with heart failure. Cochrane Database Syst Rev. 2019 Jan 29;1(1):CD003331. doi: 10.1002/14651858.CD003331.pub5. PMID 30695817
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Morris BA, Sinaei R, Smart NA. Resistance is not futile: a systematic review of the benefits, mechanisms and safety of resistance training in people with heart failure. Heart Fail Rev. 2024 Jul;29(4):827-839. doi: 10.1007/s10741-024-10402-0. Epub 2024 Apr 15. PMID 38619757
- [Background] Murray J, Bennett H, Bezak E, Perry R, Boyle T. The effect of exercise on left ventricular global longitudinal strain. Eur J Appl Physiol. 2022 Jun;122(6):1397-1408. doi: 10.1007/s00421-022-04931-5. Epub 2022 Mar 16. PMID 35296909
- [Background] Naderi-Boldaji V, Joukar S, Noorafshan A, Raji-Amirhasani A, Naderi-Boldaji S, Bejeshk MA. The effect of blood flow restriction along with low-intensity exercise on cardiac structure and function in aging rat: Role of angiogenesis. Life Sci. 2018 Sep 15;209:202-209. doi: 10.1016/j.lfs.2018.08.015. Epub 2018 Aug 7. PMID 30096385
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Russell K, Eriksen M, Aaberge L, Wilhelmsen N, Skulstad H, Remme EW, Haugaa KH, Opdahl A, Fjeld JG, Gjesdal O, Edvardsen T, Smiseth OA. A novel clinical method for quantification of regional left ventricular pressure-strain loop area: a non-invasive index of myocardial work. Eur Heart J. 2012 Mar;33(6):724-33. doi: 10.1093/eurheartj/ehs016. Epub 2012 Feb 6. PMID 22315346
- [Background] Tanaka Y, Takarada Y. The impact of aerobic exercise training with vascular occlusion in patients with chronic heart failure. ESC Heart Fail. 2018 Aug;5(4):586-591. doi: 10.1002/ehf2.12285. Epub 2018 Mar 25. PMID 29575708
- [Background] Trachsel LD, David LP, Gayda M, Henri C, Hayami D, Thorin-Trescases N, Thorin E, Blain MA, Cossette M, Lalonge J, Juneau M, Nigam A. The impact of high-intensity interval training on ventricular remodeling in patients with a recent acute myocardial infarction-A randomized training intervention pilot study. Clin Cardiol. 2019 Dec;42(12):1222-1231. doi: 10.1002/clc.23277. Epub 2019 Oct 10. PMID 31599994
- [Background] Voigt JU, Pedrizzetti G, Lysyansky P, Marwick TH, Houle H, Baumann R, Pedri S, Ito Y, Abe Y, Metz S, Song JH, Hamilton J, Sengupta PP, Kolias TJ, d'Hooge J, Aurigemma GP, Thomas JD, Badano LP. Definitions for a common standard for 2D speckle tracking echocardiography: consensus document of the EACVI/ASE/Industry Task Force to standardize deformation imaging. J Am Soc Echocardiogr. 2015 Feb;28(2):183-93. doi: 10.1016/j.echo.2014.11.003. PMID 25623220
- [Background] Caminiti G, Volterrani M, Iellamo F, Marazzi G, Manzi V, D'Antoni V, Vadala S, Di Biasio D, Catena M, Morsella V, Perrone MA. Changes in left atrial function following two regimens of combined exercise training in patients with ischemic cardiomyopathy: a pilot study. Front Cardiovasc Med. 2024 May 7;11:1377958. doi: 10.3389/fcvm.2024.1377958. eCollection 2024. PMID 38774661
- [Background] Wu P, Liu Y. The Clinical Effects of Pharmacotherapy Combined with Blood Flow Restriction and Isometric Exercise Training in Rehabilitating Patients with Heart Failure with Reduced Ejection Fraction. Rejuvenation Res. 2024 Feb;27(1):33-40. doi: 10.1089/rej.2023.0070. PMID 38308476
- [Background] Zhang D, Shen X, Qi X. Resting heart rate and all-cause and cardiovascular mortality in the general population: a meta-analysis. CMAJ. 2016 Feb 16;188(3):E53-E63. doi: 10.1503/cmaj.150535. Epub 2015 Nov 23. PMID 26598376